CLINICAL TRIAL: NCT01129804
Title: Network Support for Alcohol Treatment: Mechanisms and Effectiveness
Brief Title: Network Support for Alcohol Treatment 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-050; R01AA012827 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Consumption
Keywords: Alcohol dependence; Network Support; Cognitive-behavioral treatment; Relapse prevention; Consequences of drinking; Social network development
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Network Support (Experimental): Network Support treatment is aimed at helping patients change their social support network so that it supports abstinence. In this treatment patients will be encouraged to attend AA meetings and engage in other activities that would involve non-drinkers. These activities would be determined by the patient, with help from the therapist. Patients would learn about methods of avoiding drinking, making new friends, and getting enjoyment from activities other than drinking. In addition patients will learn specific skills intended to help them make new acquaintances and change their circle of friends.
  Interventions: Behavioral: Coping Skills Training
- Packaged Cognitive-Behavioral Treatment (Active Comparator): The purpose of Packaged Cognitive-Behavioral Treatment (PCBT) is to train patients in a variety of skills that they can use to keep themselves from drinking.
  Interventions: Behavioral: Coping Skills Training

INTERVENTIONS:
Behavioral: Coping Skills Training — Patients in both treatments will be taught skills to help them keep from drinking.

SUMMARY:
The Network Support project is part of an ongoing effort to improve treatment for alcohol dependent patients. The Network Support Project is designed to help patients change their social network from one that reinforces drinking behavior to one that reinforces sobriety.

160 patients will be assigned to one of two treatments. Each of the treatments will last 12 weeks. The first is a Network Support (NS) treatment designed to help patients develop new acquaintances and social networks. It is expected that alcohol dependent patients will benefit from increasing their contact with non-drinking people. This NS condition will be compared to a packaged CBT program for alcoholics (PCBT) that is designed to teach a number of skills to help people stop drinking, but does not address social networks per se.

In order to better understand what is happening to the investigators patients, the investigators will be using daily computerized telephone calls to ask about people's experiences. This will be done both before and after treatment. Patients will also be asked to participate in follow-up interviews every 3 months for 2 years following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 yo
* meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for alcohol dependence

Exclusion Criteria:

* acute medical or psychiatric problems that require inpatient treatment (e.g., acute psychosis, or suicide/homicide risk)
* reading ability below the fifth grade level
* lack of reliable transportation to the treatment site, or excessive commuting distance
* inability to understand English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Litt MD, Kadden RM, Kabela-Cormier E, Petry N. Changing network support for drinking: initial findings from the network support project. J Consult Clin Psychol. 2007 Aug;75(4):542-55. doi: 10.1037/0022-006X.75.4.542. PMID 17663609
- [Result] Litt MD, Kadden RM, Kabela-Cormier E, Petry NM. Changing network support for drinking: network support project 2-year follow-up. J Consult Clin Psychol. 2009 Apr;77(2):229-42. doi: 10.1037/a0015252. PMID 19309183
- [Derived] Litt MD, Kadden RM, Tennen H. Treatment response and non-response in CBT and Network Support for alcohol disorders: targeted mechanisms and common factors. Addiction. 2018 Aug;113(8):1407-1417. doi: 10.1111/add.14224. Epub 2018 Apr 20. PMID 29575339
- [Derived] Litt MD, Kadden RM, Tennen H, Kabela-Cormier E. Network Support II: Randomized controlled trial of Network Support treatment and cognitive behavioral therapy for alcohol use disorder. Drug Alcohol Depend. 2016 Aug 1;165:203-12. doi: 10.1016/j.drugalcdep.2016.06.010. Epub 2016 Jun 18. PMID 27354234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Network Support | Packaged Cognitive-Behavioral Treatment
Started | 96 | 97
Completed | 64 | 66
Not Completed | 32 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Network Support | Packaged Cognitive-Behavioral Treatment | Total
Number analyzed (Participants) | 96 | 97 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 97 | 193
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.2) | 45.1 (9.8) | 46.01 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 59 | 68 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 93 | 94 | 187
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 92 | 93 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 96 | 97 | 193

OUTCOME MEASURES:

1. Primary Outcome: Proportion Days Abstinent (PDA)
Description: PDA is based on data collected in each 90-day timeline follow-back assessment of daily drinking. PDA is calculated as the number of days out of 90 in which the patient reported 0 drinks.
Time Frame: Every 3 months out to 2 years
Population: Men and women aged 18-65 diagnosed with alcohol use disorder, moderate to severe.
Measure: Mean (Standard Deviation); unit: proportion of days abstinent
Arm/Group | Network Support | Packaged Cognitive-Behavioral Treatment
Number analyzed (Participants) | 96 | 97
proportion of days abstinent | .67 (.33) | .73 (.33)
Statistical Analysis 1: Comparison: Network Support vs Packaged Cognitive-Behavioral Treatment; Test type: Superiority — Longitudinal Linear mixed modeling; p < .04, Mixed Models Analysis — Tested the null hypothesis that slopes of PDA over time would not differ between treatment conditions, as indicated by the significance of the Treatment main effect and Treatment X Time interaction effect, at the level of p < .05; Slope = 0.1; Multilevel longitudinal modeling (MLM) with random effects and maximum likelihood estimation (Proc MIXED; SAS Institute, 1999) was used to evaluate the effects of treatment over time for each of the continuously scaled outcome variables described above. The MLM approach was used because it employs maximum likelihood estimation of covariance matrices rather than raw data, allowing us to take advantage of all data collected for anyone randomized to treatment. Each repeated dependent variable was analyzed as a unction of treatment condition, time since intake (in months), and the interaction of treatment condition by time

2. Secondary Outcome: Social Network Change
Description: Network Support for Abstinence. Minimum score=0; Maximum score =1. Higher scores indicate greater support for abstinence.
Time Frame: assessed every 6 months out to 2 years, mean change over 2 years reported
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Network Support | Packaged Cognitive-Behavioral Treatment
Number analyzed (Participants) | 96 | 97
score on a scale | .35 (.05) | .30 (.05)

ADVERSE EVENTS:
Time Frame: 27 months
Arm/Group | Network Support | Packaged Cognitive-Behavioral Treatment
All-Cause Mortality (participants affected / at risk) | 2/96 | 2/97
Serious Adverse Events (participants affected / at risk) | 30/96 | 35/97
Other Adverse Events (participants affected / at risk) | 5/96 | 5/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Network Support (N=96) | Packaged Cognitive-Behavioral Treatment (N=97)
Increased drinking from baseline (Nervous system disorders) | 30 (30) | 35 (35)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Network Support (N=96) | Packaged Cognitive-Behavioral Treatment (N=97)
Suicidal Ideation (Psychiatric disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No